CLINICAL TRIAL: NCT01962025
Title: Vanguard Multi-Centre Feasibility Trial to Determine if Buttonhole Versus Step Ladder Cannulation for High Dose Hemodialysis is Associated With Reduced Overall Cost
Brief Title: Buttonhole Versus Step Ladder Cannulation in High Dose Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20130148
Record Dates: First submitted 2013-09-16; First posted 2013-10-14 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Renal Failure
Keywords: Renal failure; Hemodialysis; Canulation technique; Training time; Cost; Patient discomfort with cannulation technique
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buttonhole needling technique (Active Comparator): the intervention is the Buttonhole needling technique for home hemodialysis
  Interventions: Procedure: Buttonhole needling technique
- Step Ladder Group (No Intervention): Patients will use step ladder needling technique

INTERVENTIONS:
Procedure: Buttonhole needling technique — the intervention is the type of needling used for home hemodialysis patients. They will be randomized to either buttonhole cannulation or stepladder cannulation
  Other Names: Buttonhole canulation in home hemodialysis patients
  Arms: Buttonhole needling technique

SUMMARY:
The purpose of the pilot study is to determine: 1) Will patients agree to be randomized to two different methods of putting needles in their arteriovenous fistula and, 2) if we can adequately coordinate all of the sites to get useful multicentre trial data

DETAILED DESCRIPTION:
To determine the feasibility of 1) randomizing patients to step-ladder versus buttonhole cannulation techniques, and 2) coordinating the multiple Canadian sites that are required for the definitive study.

Secondary Objectives: To determine 1) if buttonhole cannulation, compared to step-ladder cannulation is associated with reduced training time for high dose home hemodialysis patients, 2) if buttonhole cannulation, compared to step-ladder cannulation is associated with reduced overall cost, 3) if buttonhole cannulation, compared to step-ladder cannulation is associated with reduced complications (infection - local and systemic, radiologic/surgical interventions, re-trains for needle insertion difficulties, hematoma formation, aneurysm formation, missed insertions), and 4) if buttonhole cannulation, compared to step-ladder cannulation is associated with reduced patient discomfort with needling for intensive home hemodialysis patients

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients > 18 years old,
2. Training for home hemodialysis
3. Able to give informed consent,
4. Arteriovenous fistula 5. Life expectancy of greater than 12 months.

Exclusion Criteria:

1. Potential to be lost from the program within 12 months of training (planned living donor transplant, transfer to peritoneal dialysis (PD) or move from training centre catchment area),
2. Allergy to mupirocin,
3. Short segments or aneurysms within the arteriovenous fistula (AVF) that the attending nephrologist believes require buttonhole cannulation.,
4. Mechanical heart valves,
5. Patients who require intradermal lidocaine for needle insertion -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2017-11 (Actual); Study Completion 2019-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Zimmerman, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (3):
- Canada (3):
  - Foothills Hospital, Calgary, Alberta
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Buttonhole Needling Technique: The intervention is the Buttonhole needling technique for home hemodialysis
  Buttonhole needling technique: the intervention is the type of needling used for home hemodialysis patients. They will be randomized to either buttonhole cannulation or stepladder cannulation
  In the buttonhole technique, a constant site is used for needle placement that ultimately results in a fibrous tract. Once the tract has formed blunt needles can be used instead of sharp needles for each treatment. The presence of a tract may simplify the needle insertion technique and lead to enhanced patient confidence with needle placement.
- Step Ladder Group: Patients will use step ladder needling technique (i.e., sites will be rotated with needles placed at least 2-3cms between needle tips).
Period: Overall Study
Arm/Group | Buttonhole Needling Technique | Step Ladder Group
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Buttonhole Needling Technique: The intervention is the Buttonhole needling technique for home hemodialysis.
  Buttonhole needling technique: the intervention is the type of needling used for home hemodialysis patients. They will be randomized to either buttonhole cannulation or stepladder cannulation.
  In the buttonhole technique, a constant site is used for needle placement that ultimately results in a fibrous tract. Once the tract has formed blunt needles can be used instead of sharp needles for each treatment. The presence of a tract may simplify the needle insertion technique and lead to enhanced patient confidence with needle placement.
- Step Ladder Group: Patients will use step ladder needling technique (i.e., sites will be rotated with needles placed at least 2-3 cms between needle tips).
- Total: Total of all reporting groups
Arm/Group | Buttonhole Needling Technique | Step Ladder Group | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (13.6) | 50.8 (16.0) | 50.4 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 7 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 5 | 11
  Asian | 1 | 1 | 2
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 6 | 14
Etiology renal disease [Count of Participants; unit: Participants]
  Diabetes mellitus | 3 | 1 | 4
  Polycystic kidney disease | 0 | 0 | 0
  Glomerulonephritis | 0 | 1 | 1
  Other | 5 | 4 | 9
End Stage Renal Disease (ESRD) Vintage [Mean (Standard Deviation); unit: years] — The duration of time between the first day of dialysis treatment and the day of kidney transplantation.
  years | 8.0 (11.1) | 6.0 (6.1) | 6.7 (9.7)
Previous access [Number; unit: participants]
  Had 1 Central Venous Catheter (CVC) | 2 | 1 | 3
  Had >1 CVC | 4 | 3 | 7
  No CVC | 1 | 2 | 3
  Had 1 Arteriovenous Fistula or Graft (AVF/AVG) | 2 | 0 | 2
  Had 1+ AVF/AVG | 0 | 1 | 1
  No AVF/AVG | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Participant Recruitment and Site Coordination
Description: The percent of qualified patients enrolled in the study for the pilot study to be successful will be ≥70%. If we can not reach this target we will not move forward with the definitive study. The pilot study will also allow us to see if we can coordinate multiple sites in needling techniques and determine if we can move forward with the definitive study.
Time Frame: 2 years
Population: Intent to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Buttonhole Needling Technique | Step Ladder Group
Number analyzed (Participants) | 8 | 6
Participants | 8 | 6

2. Secondary Outcome: Participant Training Time
Description: Time in Days that it takes to train participants to perform home hemodialysis (document time in days from start of training until discharge home to do self-care). Unit of measure is number of days required to independently perform home hemodialysis
Time Frame: Up to 90 days
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Buttonhole Needling Technique | Step Ladder Group
Number analyzed (Participants) | 8 | 6
days | 19 (5) | 29 (14)

3. Secondary Outcome: Cost
Description: Will incorporate the cost of training and complications
Time Frame: 12 Months
Population: No formal costing information was collected as the data linkages were not established for the feasibility trial period.
Arm/Group | Buttonhole Needling Technique | Step Ladder Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Complications
Description: To determine whether buttonhole cannulation, compared to step-ladder cannulation, is associated with reduced complications (infection - local and systemic, radiologic/surgical interventions, re-trains for needle insertion difficulties, hematoma formation, aneurysm formation, missed insertions).
Time Frame: 12 Months
Population: Intent to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Buttonhole Needling Technique | Step Ladder Group
Number analyzed (Participants) | 8 | 6
Participants
  Contact dermatitis | 3 | 1
  Stenosis Requiring Angioplasty | 4 | 3
  Aneurysm | 3 | 0
  Hematoma | 1 | 5
  Infection - local and systemic | 0 | 0
  Radiologic/surgical interventions | 2 | 0
  Re-training for needle insertion difficulties | 0 | 0
  Missed insertions | 8 | 6

5. Secondary Outcome: Pain With Needling
Description: Pain/discomfort during cannulation will be measured using a 10cm (0 mm to 100 mm) visual analogue scale, which ranges from "No Pain" (0 mm) on the left side to "Extreme Pain" (100 mm) on the right. The participant is instructed to place a mark on the scale according to the amount of pain felt during needling the fistula that day. The visual analogue scale with be completed at baseline, end of training, and 2 months after graduating training. The mean of these three assessments will be calculated.
Time Frame: baseline, end of training (2 months), and 2 months after graduating training (4 months)
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Buttonhole Needling Technique | Step Ladder Group
Number analyzed (Participants) | 8 | 6
mm | 17.4 (25.1) | 10.7 (7.9)

ADVERSE EVENTS:
Time Frame: During study period - at start, 6 months and at completion of study (12 months).
Arm/Group | Buttonhole Needling Technique | Step Ladder Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT01962025/Prot_SAP_000.pdf